CLINICAL TRIAL: NCT04475146
Title: Impact de la Visualisation d'Une vidéo Explicative Sur la qualité de la préparation Intestinale
Brief Title: Impact of Visualisation an Explanatory Video on the Quality of Bowel Preparation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PREPAVIDEO
Record Dates: First submitted 2020-07-02; First posted 2020-07-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colonoscopy
Keywords: video of bowel preparation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard information and video visualization: Standard information and video visualization
  Interventions: Other: video vizualisation
- Standard information, no video: Standard information, no video

INTERVENTIONS:
Other: video vizualisation — video vizualisation
  Groups: Standard information and video visualization

SUMMARY:
The research hypothesis is that video visualization improves the quality of bowel preparation and the patients' understanding of the modalities of bowel preparation.

DETAILED DESCRIPTION:
The prescription of colonoscopy is performed by a gastroenterologist, who chooses the type of bowel preparation. During this consultation, the doctor explains to the patient the bowel preparation, then gives the patient the prescription with the type of product and a sheet explaining the diet without residues.

The time between this consultation and the colonoscopy is sometimes long. The idea of this study is to accompany this information on intestinal preparation with a video that details the different stages of intestinal preparation by MOVIPREP. Indeed, studies have in the past shown an improvement in the quality of intestinal preparation with the help of better information to patients (educational booklet, or smartphone application)

ELIGIBILITY:
Inclusion Criteria

* Major patient
* Patient with first indication of colonoscopy
* Colonoscopy performed in outpatient with preparation by MOVIPREP
* Patient affiliated with Social Security
* Informed consent signed by the patient

Exclusion Criteria:

* Hospitalized patients
* With no Internet access, or no access to the email
* Blind patients
* Patient who don't speak French
* Pregnant woman
* Severe constipation (3 stools/week) or long-term laxatives
* History of partial or total colectomy
* Other preparation product

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patients, without legal protection measures, understanding French and having access to the internet and an email address. Patient having a first outpatient colonoscopy with preparation by MOVIPREP.
  The study will be proposed by the investigator to patients followed for colonoscopy in the department of Hepato-gastroenterology. If patients accepted to participate in the protocol and the informed consent form is signed, patients will be included in the protocol.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of colonoscopy percentage with a Boston score of 7 or higher and a score of 2 or higher in each segment, in group 1 "standard information and video visualization" versus in group 2 "standard information." | Immediately after the colonoscopy
  Boston score

SECONDARY OUTCOMES:
A scale of understanding and satisfaction in relation to the quality of Information on intestinal preparation. | 2 hours after the colonoscopy
  Satisfaction and Understanding Questionnaires (Likert Scale)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre hospitalier intercommunal de Créteil, Créteil
  - CHI Villeneuve St George, Villeneuve-Saint-Georges